CLINICAL TRIAL: NCT06961643
Title: Investigation of Pharmacokinetics and Safety of HRS-7535 in Subjects With Mild and Moderate Hepatic Impairment and Normal Hepatic Function
Brief Title: Investigation of Pharmacokinetics and Safety of HRS-7535 in Subjects With Hepatic Impairment and Normal Hepatic Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7535-109
Record Dates: First submitted 2025-05-06; First posted 2025-05-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): Subjects with mild hepatic impairment.
  Interventions: Drug: HRS-7535 Tables
- Treatment group B (Experimental): Subjects with moderate hepatic impairment.
  Interventions: Drug: HRS-7535 Tables
- Treatment group C (Experimental): Subjects with normal hepatic function.
  Interventions: Drug: HRS-7535 Tables

INTERVENTIONS:
Drug: HRS-7535 Tables — Oral HRS-7535 tables.

SUMMARY:
The study is being conducted to compare the pharmacokinetics and safety of HRS-7535 in subjects with mild to moderate hepatic impairment and normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study procedures and methods, participate voluntarily and be able to complete the study according to the protocol requirements, and sign the informed consent form (ICF) in writing.
2. Aged 18-70 years old on the date of signing the ICF (including the threshold), both male and female.
3. At the time of screening, male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg; body mass index (BMI): 18~32 kg/m2 (including the threshold).

Exclusion Criteria:

1. In the judgment of the investigator, may be allergic to the study drug or its components.
2. Smoking an average of more than 10 cigarettes per day within 3 months prior to screening.
3. Alcoholics of within 3 months prior to screening, who consume more than 14 units of alcohol per week (1 unit=beer)360 mL of alcohol, or 45 mL of strong liquor with an alcohol content of 40%, or 150 mL of wine.
4. History of drug or substance abuse, or a positive urine drug test at screening.
5. Donated or lost ≥ 400 mL of blood within 3 months prior to screening.
6. Individuals with a history of severe hypoglycemia.
7. Undergone surgery within 6 months prior to screening, or plan to undergo surgery during the trial period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration of HRS-7535 (Cmax) | Post-dose at day 1 to day 4.
Area under the concentration curve from time 0 to the last quantifiable concentration (AUC0-t) | Post-dose at day 1 to day 4.
Area under the concentration curve from time 0 to extrapolated infinite time (AUC0-inf) | Post-dose at day 1 to day 4.

SECONDARY OUTCOMES:
Time to maximum plasma concentration (Tmax) | Post-dose at day 1 to day 4.
Terminal half-life (t1/2) | Post-dose at day 1 to day 4.
Apparent clearance (CL/F) | Post-dose at day 1 to day 4.
Apparent volume of distribution (Vz/F) | Post-dose at day 1 to day 4.
Adverse events (AEs) | Screening period up to Day 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Infectious Disease Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided